CLINICAL TRIAL: NCT03466827
Title: A Phase II Study of Selinexor (KPT-330) in Patients With Advanced Thymic Epithelial Tumour (TET) Progressing After Primary Chemotherapy.
Brief Title: Selinexor in Patients With Advanced Thymoma and Thymic Carcinoma
Acronym: TET-SEL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Morten Mau-Soerensen (Other)
Collaborators: Institut Curie (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other); Hospices Civils de Lyon (Other); GSO Global Clinical Research BV (Other); Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor-Investigator, Morten Mau-Soerensen, Chief Physician, MD, PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TET-SEL
Record Dates: First submitted 2018-03-09; First posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Thymoma; Advanced Thymic Epithelial Tumour
MeSH Terms: conditions — Thymoma | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Selinexor — Selinexor 60 mg oral tablets will be administered twice weekly, either Monday/Wednesday or on Tuesday/Thursday or on Wednesday/Friday in a 3-weeks-on and 1-week-off Schedule.
  Other Names: KPT-330

SUMMARY:
The aim of the study is to determine the efficacy of selinexor in adults with TETs determined by overall response rate (RECIST 1.1) in two parallel cohorts of patients with advanced thymomas or thymic carcinomas. The study is an international, multicenter, open label phase II trial using Simons two stage design. The study population is adults with histologically confirmed, advanced, inoperable TETs who are progressing after treatment with least one platinum containing chemotherapy regimen.

This study is comprised of 2 similar phase II tirals, one running in EU (25 patients) and one running in US (25 patients).

There are two study arms:

Arm A: Thymoma

* Stage 1: 15 patients
* Stage 2: 10 patients

Arm B: Thymic carcinoma

* Stage 1: 15 patients
* Stage 2: 10 patients

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced TET (thymoma or thymic carcinoma)
* Inoperable per local Investigator (Masaoka Stage III or IV)
* Progression after treatment with least one platinum containing chemotherapyregimen
* Measurable disease (RECIST 1.1)
* Age ≥18 years
* ECOG PS <2
* Patients must have recovered from the toxic effects of prior therapy at the time of initiation of the study drug unless toxicity is stable.
* A 4 weeks interval from any investigational agents or cytotoxic chemotherapy to start of study is required
* Signed informed consent
* Adequate bone marrow function and organ function:

  * Hematopoietic function: total white blood cell count (WBC) ≥ 3000/mm³, absolute neutrophil count (ANC) ≥ 1500/mm³, platelet count ≥ 100,000/mm²
  * Hepatic function: bilirubin < 1.5 times the upper limit of normal (ULN), ALT < 2.5 times ULN or ALT < 5.0 times ULN in the presence of liver metastases
  * Creatinine clearance > 30 ml/min according to Cockcroft-Gault
* Patients of childbearing potential must agree to use adequate birth control during and for 3 months after participation in this study

Exclusion Criteria:

* No significant medical illness that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy, including

  * Unstable cardiovascular function
  * Known active hepatitis A, B, or C infection; or known to be positive for HCV RNA or HBsAg (HBV surface antigen)
  * Markedly decreased visual acuity
  * Active infection requiring intravenous antibiotics
* Pregnancy or breast-feeding
* Symptomatic brain metastasis requiring corticosteroids
* Uncontrolled autoimmune disorders. Patients with autoimmune disorders under control on medication may be included. Patients with pure red cell aplasia may be included if haemoglobin levels are relatively stable on transfusions or medication
* Any other cancer (excluding radically operated localised squamous skin cancer) with clinical activity within the last 2 years
* Significantly diseased or obstructed gastrointestinal tract, malabsorption, uncontrolled vomiting or diarrhea or inability to swallow oral medications
* No dehydration of NCI-CTCAE grade ≥ 1
* Serious psychiatric or medical conditions that could interfere with treatment.
* No history of organ allograft
* No concurrent therapy with approved or investigational anticancer therapeutics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-10-12 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 24 months
  To determine the overall response rate according to RECIST 1.1

SECONDARY OUTCOMES:
Progression Free Survival | 6 months
  To determine six months progression free survival of patients with TET treated with selinexor
Adverse Events | 24 months
  The number of adverse events as determined by Common Terminology Criteria for Adverse Events (CTCAEs) version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Morten Mau-Soerensen, MD, PhD, Study Director — Rigshospitalet, Denmark
Locations (4):
- Rigshospitalet, Copenhagen, Denmark
- France (3):
  - Hospices Civils de Lyon, Lyon
  - Intitut Curie, Paris
  - Intitut Gustave Roussy, Paris

IPD SHARING:
Plan to Share IPD: No